CLINICAL TRIAL: NCT01046903
Title: An Observational Study On The Safety And Tolerability Of Prolonged Thrombosis Prophylaxis With Fragmin® (Dalteparin Sodium) In Patients Undergoing Major Orthopedic Surgery
Brief Title: An Observational Study On The Safety And Tolerability Of Prolonged Thrombosis Prophylaxis With Fragmin®
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6301085
Record Dates: First submitted 2010-01-04; First posted 2010-01-12 (Estimated); Results first posted 2012-02-13 (Estimated); Last update posted 2012-02-27 (Estimated); Status verified 2012-02

CONDITIONS: Venous Thromboembolism
Keywords: observational prolonged thromboprophylaxis
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dalteparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Fragmin® (Dalteparin Sodium)

INTERVENTIONS:
Drug: Fragmin® (Dalteparin Sodium) — Administered per prescribing physician

SUMMARY:
The objective of this study is to observe the safety, tolerability, and compliance in the use of Fragmin® for prolonged thromboprophylaxis in post-surgery high-risk orthopedic patients.

DETAILED DESCRIPTION:
All patients prescribed Fragmin® (Dalteparin Sodium) for prolonged thromboprophylaxis will be eligible for study

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, undergoing major orthopedic surgery
* At least 18 years old

Exclusion Criteria:

* Hypersensitivity to Fragmin or other low molecular weight heparins or unfractioned heparin;
* History of heparin induced thrombocytopaenia type II
* Acute gastroduodenal ulcer, cerebral haemorrhage, or other active haemorrhage.
* Serious coagulation disorder;
* Septic endocarditis;
* Injuries to and operations in the central nervous system, eye and ear within one month before orthopaedic surgery;
* Spinal or epidural anesthesia or other procedures requiring spinal puncture and concomitant treatment with high doses of dalteparin (such as those needed to treat acute deep vein thrombosis, pulmonary embolism, and Unstable coronary artery disease);
* Patients with serum creatinine level > 150 umol/l;
* Platelet count of less than 100 000 per cubic millimeter at the beginning of the therapy;
* High probability that patient will not return to the centre for follow-up;
* Patient on oral anticoagulation therapy in the last 7 days;
* Ongoing anticoagulant therapy with other medications or non-pharmacologic therapy during the study period;
* Weight less than 40 kg;
* Simultaneous participation in another pharmacological study or receiving any investigational drug 30 days or less before surgery;
* Pregnancy or breastfeeding;
* Clinically significant hepatic dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The adult population (women and men) after major orthopedic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6301085&StudyName=An%20Observational%20Study%20On%20The%20Safety%20And%20Tolerability%20Of%20Prolonged%20Thrombosis%20Prophylaxis%20With%20Fragmin%AE%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Dalteparin Sodium: Dalteparin Sodium (Fragmin) 2500 International Unit (IU)/0.2 milliliter (mL) and 5000 IU/2 mL subcutaneously (s.c) as per registered indications for 5 weeks.
Period: Overall Study
Arm/Group | Dalteparin Sodium
Started | 503
Completed | 475
Not Completed | 28
Not completed — Lost to Follow-up | 16
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 3
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Groups:
- Dalteparin Sodium: Dalteparin Sodium (Fragmin) 2500 IU/0.2 mL and 5000 IU/2 mL s.c as per registered indications for 5 weeks.
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Age Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 340
  Male | 163
Primary diagnosis [Number; unit: Participants] | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Medical history [Number; unit: Participants] | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Procedures After Primary Diagnosis [Number; unit: Participants] | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Thromboembolic Disease Assessment [Number; unit: Participants] — Thromboembolism is the formation of blood clot in the blood vessels due to an embolus (a detached intravascular mass capable of clogging arterial capillary beds at a site far from its origin).Thromboembolic disease was assessed based on clinical examination only (presence of symptoms).
  Participants | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Prior Surgery History [Number; unit: Participants] | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Prior Study Medications [Number; unit: Participants] | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.
Concomitant Study Medications [Number; unit: Participants] | NA — Data for this pre-specified outcome measure was collected and reported in individual participant listings but not statistically summarized for analysis.

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Participant's Dosage Regimen
Description: Approved dosage regimens for Fragmin in major orthopedic surgery included; (1): first dose of Fragmin 5000 IU in the evening before the day of surgery, followed by daily doses of 5000 IU up to 5 weeks; (2): first dose of Fragmin 2500 IU 2 hours before surgery, and a second dose of 2500 IU 8 to 12 hours later, not earlier than 4 hours after surgery, followed by daily doses of 5000 IU up to 5 weeks or (3): first dose of Fragmin 2500 IU 4 to 8 hours postoperatively, followed by daily doses of 5000 IU up to 5 weeks.
Time Frame: Baseline up to Week 5
Population: The Safety Analysis Set included all those participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Participants
  Dosage Regimen 1 | 327
  Dosage Regimen 2 | 2
  Dosage Regimen 3 | 115
  Other | 59

2. Other Pre Specified Outcome: Number of Participants With Risk Factors
Description: Risk factors evaluated for vascular thromboembolism (VTE) were age (above 40 years, but age was not a strong risk factor as a prediction of potential VTE episode), gender (primarily females but males after 65 years also influenced VTE episode), obesity, pregnancy, liver disease, kidney disease, hormone therapy, immobilization, previous surgery, concomitant malignant disease, positive family history, varicose veins, smoking, chemotherapy, catheter in vein, Heart Failure III New York Heart Association (NYHA) and Heart Failure IV NYHA.
Time Frame: Baseline
Population: The Safety Analysis Set included all those participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Participants
  Age | 353
  Obesity | 205
  Gender | 291
  Pregnancy | 12
  Liver disease | 8
  Kidney disease | 7
  Hormone therapy | 20
  Immobilization | 51
  Previous surgery | 257
  Concomitant malignant disease | 11
  Positive family history | 16
  Varicose veins | 181
  Smoking | 92
  Chemotherapy | 4
  Catheter in vein | 204
  Heart failure III New York Heart Association(NYHA) | 6
  Heart failure IV NYHA | 0

3. Other Pre Specified Outcome: Number of Participants With Thromboembolism
Description: Thromboembolism is the formation of blood clot in the blood vessels due to an embolus (a detached intravascular mass capable of clogging arterial capillary beds at a site far from its origin).
Time Frame: Baseline up to Week 5
Population: The Safety Analysis Set included all those participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Participants | 3

4. Other Pre Specified Outcome: Number of Participants With Bleeding
Description: Major bleeding: defined as fatal bleeding, clinically overt bleeding causing a fall in hemoglobin more than or equal to 20 gram/litre (g/L) (2 g/decilitre [dL]), clinically overt bleeding leading to transfusion of more than or equal to 2 units of whole blood or red cells, or symptomatic bleeding in areas of special concern (intracranial, retroperitoneal, intraocular, intraspinal, pericardial, intramuscular with compartmental syndrome, or intraarticular). Minor bleeding was defined as bleeding that did not meet the definition of major bleeding.
Time Frame: Baseline up to Week 5
Population: The Safety Analysis Set included all those participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Participants
  Major Bleeding | 0
  Minor Bleeding | 0

5. Other Pre Specified Outcome: Participant's Global Evaluation of Treatment
Description: Participant's global evaluation of treatment for overall response and comfort was evaluated on the four point categorical scale: excellent, good, fair and poor.
Time Frame: Baseline up to Week 5
Population: The Safety Analysis Set included all those participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Participants
  Overall response (Excellent) | 236
  Overall response (Good) | 220
  Overall response (Fair) | 20
  Overall response (Poor) | 1
  Overall comfort (Excellent) | 129
  Overall comfort (Good) | 238
  Overall comfort (Fair) | 106
  Overall comfort (Poor) | 4

6. Other Pre Specified Outcome: Physician's Assessment of Tolerability of Treatment
Description: Tolerability of treatment as assessed by physician was evaluated on the five point categorical scale: excellent, very good, good, fair, poor.
Time Frame: Baseline up to Week 5
Population: The Safety Analysis Set included all those participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Participants
  Excellent | 354
  Very good | 116
  Good | 10
  Fair | 0
  Poor | 0
  Not reported | 23

7. Primary Outcome: Physician's Assessment of Efficacy of Treatment
Description: Efficacy of treatment as assessed by physician was evaluated on the 5 point categorical scale: excellent, very good, good, fair, poor.
Time Frame: Baseline up to Week 5
Population: The Full Analysis Set (FAS) included all those participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Participants
  Excellent | 432
  Very good | 44
  Good | 2
  Fair | 2
  Poor | 1
  Not reported | 22

8. Other Pre Specified Outcome: Administration Schedule of Treatment
Description: Administration schedule for Fragmin in major orthopedic surgery Included was categorized as; (1): first dose of Fragmin 5000 IU in the evening before the day of surgery, followed by daily doses of 5000 IU up to 5 weeks; (2): first dose of Fragmin 2500 IU 2 hours before surgery, and a second dose of 2500 IU 8 to 12 hours later, not earlier than 4 hours after surgery, followed by daily doses of 5000 IU up to 5 weeks or (3): first dose of Fragmin 2500 IU 4 to 8 hours postoperatively, followed by daily doses of 5000 IU up to 5 weeks.
Time Frame: Baseline up to Week 5
Population: The Safety Analysis Set included all those participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Participants
  Administration Schedule 1 | 327
  Administration Schedule 2 | 2
  Administration Schedule 3 | 115
  Other | 59

9. Other Pre Specified Outcome: Number of Participants Compliant With the Treatment
Description: Compliance was defined as participants documented with Dalteparin Sodium up to 5 weeks after initiation of thromboprophylaxis.
Time Frame: Baseline up to Week 5
Population: Data was collected but not statistically summarized for analysis.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Number of Participants With Hematoma
Description: Hematoma is a localized collection of blood outside of a blood vessel. It includes subcutaneous hematoma and injection-site hematoma.
Time Frame: Baseline up to Week 5
Population: The Safety Analysis Set included all those participants who received at least 1 dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Dalteparin Sodium
Number analyzed (Participants) | 503
Participants | 2

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Dalteparin Sodium
Serious Adverse Events (participants affected / at risk) | 26/503
Other Adverse Events (participants affected / at risk) | 46/503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin Sodium (N=503)
Acute coronary syndrome (Cardiac disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 2
Device dislocation (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Postoperative wound infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Periprosthetic fracture (Injury, poisoning and procedural complications) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 4
Paralysis (Nervous system disorders) | 1
Sciatic nerve palsy (Nervous system disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Skin sensitisation (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 3
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalteparin Sodium (N=503)
Anaemia (Blood and lymphatic system disorders) | 5
Arrhythmia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 7
Device dislocation (General disorders) | 1
Injection site haematoma (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 1
Soft tissue inflammation (General disorders) | 1
Asymptomatic bacteriuria (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1
Anaesthetic complication (Injury, poisoning and procedural complications) | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1
Post procedural oedema (Injury, poisoning and procedural complications) | 1
Procedural vomiting (Injury, poisoning and procedural complications) | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1
Gout (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Hypotonia (Nervous system disorders) | 1
Anxiety disorder (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 5
Sleep disorder (Psychiatric disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 5
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 2
Venous thrombosis limb (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.